CLINICAL TRIAL: NCT06936644
Title: A Multicenter, Single-arm Phase II Study to Evaluate the Efficacy and Safety of Fulzerasib (IBI351) in Combination With Ivonescimab (AK-112) in First-line Treatment of Advanced or Metastatic Non-small Cell Lung Cancer Patients With KRAS G12C Mutation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Innovent Biologics, Inc. (Other); Akesobio (Industry)
Responsible Party: Principal Investigator, Zhong Runbo, The chief physician of pneumology department, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI351IIS006
Record Dates: First submitted 2025-04-14; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: KRAS G12C Lung Cancer

STUDY DESIGN:
Intervention Model Description: the combination of IBI351 plus AK112
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The combination of IBI351 plus AK112 (Experimental)
  Interventions: Drug: IBI351+AK112

INTERVENTIONS:
Drug: IBI351+AK112 — The advanced or metastatic non-small cell lung cancer patients with KRAS G12C mutation will receive the combination of fulzerasib (IBI351) with ivonescimab (AK-112) in first-line treatment
  Other Names: fulzerasib; ivonescimab

SUMMARY:
A multicenter, single-arm Phase II study to evaluate the efficacy and safety of fulzerasib (IBI351) in combination with ivonescimab (AK-112) in first-line treatment of advanced or metastatic non-small cell lung cancer patients with KRAS G12C mutation

ELIGIBILITY:
Inclusion Criteria:

1. Sign the Informed Consent Form (ICF) and be able to comply with the visit and related procedures as stipulated in the protocol.
2. Be male or female, aged ≥18 and ≤75 years old.
3. Have an expected survival time of ≥6 months.
4. Have histologically or cytologically confirmed locally advanced (IIIB/IIIC stage), metastatic or recurrent (IV stage) non-small cell lung cancer (NSCLC) that is not operable and not suitable for radical concurrent chemoradiotherapy, as classified by the 8th edition of the TNM staging system of the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer.
5. All subjects must have a written test report before enrollment to prove the presence of KRAS G12C mutation; and must have no sensitive mutations of Epidermal Growth Factor Receptor (EGFR), Anaplastic Lymphoma Kinase (ALK), or other gene mutation types approved by the National Medical Products Administration (NMPA) for first-line treatment of NSCLC.
6. Have at least one measurable lesion according to RECIST 1.1 criteria.
7. Have not received any systemic anti-tumor treatment for locally advanced or metastatic NSCLC before; previous adjuvant therapy is allowed, but the interval between the last adjuvant therapy or last radical radiotherapy and disease recurrence should be at least 6 months.
8. Have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1.
9. Have adequate organ and bone marrow function (subjects who have received any cell or growth factor therapy within 2 weeks before the first administration of the study drug should be excluded), defined as follows:

1) Blood routine: Absolute neutrophil count (ANC) ≥1.5×109/L or within the normal range; platelet (PLT) count ≥100×109/L; hemoglobin (HGB) content ≥9.0 g/dL.

2) Liver function: Serum total bilirubin (TBIL) ≤1.5×Upper Limit of Normal Value (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN.

3) Renal function: Serum creatinine (Cr) ≤1.5×ULN or clearance of creatinine (CCr) ≥50 mL/min, calculated by the Cockcroft-Gault formula (using actual body weight); urine routine test shows urine protein <2+; for subjects with urine protein ≥2+ at baseline as detected by urine test strips, a 24-hour urine collection should be performed and the protein content in 24-hour urine should be <1 g (if both methods are used, the value obtained from 24-hour urine collection will be used to determine eligibility). 4) Coagulation function: Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN and International Normalized Ratio (INR) ≤ 1.5; 10. Female subjects of childbearing age or male subjects whose partners are of childbearing age must take effective contraceptive measures throughout the treatment period and for 180 days after the treatment.

11. Female subjects have evidence of postmenopausal status, or the urine or serum pregnancy test results of premenopausal female subjects are negative.

Exclusion Criteria:

Subjects should not be enrolled in this study if they meet any of the following criteria:

1. Histological or cytological pathology confirms the presence of small cell carcinoma, neuroendocrine carcinoma, sarcoma, lymphoepithelioma-like carcinoma, salivary gland tumors, or mesenchymal tumor components.

2. Have significant cardiovascular or cerebrovascular diseases, such as:

1. Experienced definite cardiovascular abnormal events within 6 months, such as myocardial infarction, angina pectoris, heart failure, severe arrhythmia, or undergone angioplasty, vascular stent implantation, coronary artery bypass surgery, etc.
2. Have clinically significant QT/QTcF interval prolongation (QTcF > 470ms for females or > 450ms for males).
3. Experienced definite cerebrovascular abnormal events within 3 months, such as cerebral hemorrhage or cerebral infarction.

3. Active central nervous system metastases (such as brain metastases or leptomeningeal metastases) are not eligible for enrollment. For subjects with brain metastases who have received radiotherapy or local treatment, if no hormones or antiepileptic drugs are used, they must be asymptomatic within at least 7 days after radiotherapy to be eligible for enrollment; if hormones or antiepileptic drugs are used, they must be asymptomatic within at least 7 days after drug withdrawal and the investigator deems the brain metastases to be stable, they can be eligible for enrollment; if stable brain metastases patients have not received radiotherapy or hormone or antiepileptic drug treatment, they can be eligible for enrollment after the investigator deems the brain metastases to be stable.

4. Currently have clinically significant interstitial lung disease, radiation pneumonitis, drug-related pneumonitis, active pulmonary tuberculosis, pneumoconiosis, or have ≥ grade 2 other types of pneumonia, or have severe lung function impairment confirmed by pulmonary function tests (FEV1 or DLCO or DLCO/VA < 40% of predicted values).

5. Have significant gastrointestinal diseases, such as intractable hiccups, nausea, vomiting, severe gastrointestinal ulcers, liver cirrhosis, active gastrointestinal bleeding, or other diseases that affect swallowing tablets or significantly affect the absorption of oral drugs.

6. Have major acute or chronic infections, including:

1. Active infections requiring systemic treatment;
2. Positive human immunodeficiency virus antibody (HIV-Ab) at baseline, acute or chronic active hepatitis B (defined as positive HBsAg and/or HBcAb and HBV-DNA copy number higher than 2500 copies/ml or 500IU/ml), or acute or chronic active hepatitis C (positive HCV antibody and HCV-RNA higher than the detection limit of the analytical method);
3. Active pulmonary tuberculosis. 7. Accompanied by recurrent drainage or refractory pleural or peritoneal effusion or pericardial effusion.

8. Accompanied by other poorly controlled systemic diseases, such as uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg) or diabetes despite standard treatment.

9. Have a history of significant bleeding tendency or coagulation disorders; have significant clinical bleeding symptoms within 4 weeks before enrollment, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing or expectorating ≥ 1 teaspoon of fresh blood or small blood clots or only coughing blood without sputum, subjects with blood in sputum are allowed to enroll), nasal bleeding (excluding epistaxis and retracted nasal blood); imaging studies during the screening period show that the tumor surrounds important blood vessels or has obvious necrosis or cavities, and the investigator deems that enrollment in the study would cause a bleeding risk.

10. Tumor invades or compresses surrounding important organs (such as the aorta, heart and pericardium, superior vena cava, trachea, esophagus, etc.) or has a risk of esophagotracheal fistula or esophagopleural fistula; mediastinal lymph node metastasis of the tumor invades the trachea or main bronchus. 11. Participants with other malignant tumors within 2 years before entering the study, except for appropriately treated cervical carcinoma in situ, focal cutaneous squamous cell carcinoma, basal cell carcinoma, prostate cancer that does not require treatment, ductal carcinoma in situ of the breast, and superficial non-muscle-invasive urothelial carcinoma.

12. Participants who have previously received KRAS G12C inhibitor treatment. 13. Participants who have previously received immunotherapy, including immune checkpoint inhibitors (such as anti-PD-1/L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), and any other treatments targeting tumor immune mechanisms.

14. Participants who have previously received systemic anti-angiogenic therapy, including but not limited to bevacizumab and its biosimilars, endostar, small molecule TKIs, ramucirumab, etc.

15. Participants who have received systemic treatment with traditional Chinese medicine with anti-tumor indications within 1 week before the first dose or with drugs that have immunomodulatory effects within 2 weeks before the first dose (including thymosin, interferon, interleukin, except for local use to control pleural effusion).

16. Participants who have received therapeutic or palliative radiotherapy (excluding cranial radiotherapy) or local treatment within 14 days before the first dose of this study.

17. Participants who have received chemotherapy, targeted therapy, immunotherapy, other investigational drugs or investigational devices, or other anti-tumor treatments within 28 days or 5 half-lives (whichever is shorter) before the first dose of this study.

18. Participants who have undergone surgery that may affect the administration or evaluation of this study within 28 days before enrollment (excluding biopsy).

19. Participants who have received known CYP2D6, CYP3A4, P-gp, and BCRP sensitive substrates within 14 days or 5 half-lives (whichever is longer) before the first dose of this study, and the therapeutic window of the substrate is narrow, unless agreed by the investigator and the sponsor to be enrolled.

20. Participants who are simultaneously involved in another interventional clinical study, except for observational (non-interventional) clinical studies or those in the follow-up stage after the end of an interventional study.

21. Participants who have used immunosuppressive drugs within 4 weeks before the first dose of study treatment, excluding nasal sprays, inhalation or other local routes of glucocorticoids or systemic glucocorticoids at physiological doses (i.e., no more than 10mg/day of prednisone or equivalent doses of other glucocorticoids), or glucocorticoids used to prevent contrast agent allergy.

22. Participants who have received live attenuated vaccines within 4 weeks before the first dose of study treatment or plan to receive them during the study period.

23. Note: Inactivated virus vaccines for seasonal influenza by injection are allowed within 4 weeks before the first dose of study treatment; however, live attenuated influenza vaccines are not allowed.

24. Participants with known or suspected autoimmune diseases or a history of such diseases within the past 2 years (participants with vitiligo, psoriasis, alopecia, or Graves' disease that did not require systemic treatment in the past 2 years, hypothyroidism requiring only thyroid hormone replacement therapy, and type 1 diabetes requiring only insulin replacement therapy can be enrolled).

25. Participants with active or a history of definite inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea).

26. Participants with a known history of primary immunodeficiency. 27. Participants with a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

28. Participants with a history of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolic event within 3 months before enrollment (implantable venous access ports or catheter-related thrombosis, or superficial venous thrombosis are not considered "serious" thromboembolic events).

29. Participants with known allergies to study treatment or any of its components.

30. Pregnant or lactating women. 31. Other situations that the researcher deems unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
ORR | about 6 month
  the investigator assessed objective response rate

IPD SHARING:
Plan to Share IPD: Undecided